CLINICAL TRIAL: NCT06724276
Title: Effectiveness of Combined Treatment Methods for Non-Healing Wounds in Patients with Chronic Lower Extremity Arterial Disease: a Comparative Study
Brief Title: Combined Treatment for Non-Healing Wounds in Chronic Lower Extremity Arterial Disease: a Comparative Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulip Medicine (Other)
Collaborators: National Research Oncology and Transplantology Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Azat Chinaliyev, Head of department, National Research Oncology and Transplantology Center, Kazakhstan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NROC
Record Dates: First submitted 2024-06-11; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Obliterans, Arteriosclerosis; Peripheral Arterial Disease; Diabetic Foot
Keywords: balloon angioplasty; stenting of vessels; atherosclerosis; diabetes mellitus; fibroblast
MeSH Terms: conditions — Arteriosclerosis Obliterans; Peripheral Arterial Disease; Diabetic Foot; Atherosclerosis; Diabetes Mellitus | interventions — Angioplasty, Balloon

STUDY DESIGN:
Intervention Model Description: This study will be a randomized controlled trial, adhering to the CONSORT checklist. Randomization will be conducted using the RandStuff online random number generator, where the number on the stationary card will correspond to the patient's number.
  The study will include 116 participants with long-term non-healing wounds from chronic obliterating disease of the lower extremities across three cities in Kazakhstan.
  Groups:
  * Main: 58
  * Control: 58
  * Total: 116
  * Main Group: Combined treatment (balloon angioplasty or stenting + fibroblast transplantation).
  * Control Group: Endovascular interventions + traditional debridement. Procedures will include balloon angioplasty or stenting, followed by fibroblast transplantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combined treatment (Experimental): Combined treatment (balloon angioplasty or stenting + fibroblast transplantation).
  Interventions: Procedure: balloon angioplasty and stenting of lower extremity vessels + fibroblasts
- Endovascular treatment (Active Comparator): Endovascular interventions + traditional debridement.
  Interventions: Procedure: balloon angioplasty and stenting of lower extremity vessels

INTERVENTIONS:
Procedure: balloon angioplasty and stenting of lower extremity vessels + fibroblasts — A balloon or a stent of the required size (according to the intrinsic diameter of the affected vessel) is delivered to the affected area, sequential balloon dilatation with exposure of up to 5 minutes or stenting of the vessel is performed. After completion, control angiography is performed with evaluation of the result. Instruments, introdjuncer are removed. Manual compression haemostasis (up to 20 minutes over the puncture site) followed by aseptic pressure dressing on the puncture site for 12 hours with bed rest. After surgery, fibroblasts will be applied to the wound for 24 hours.
  Arms: combined treatment
Procedure: balloon angioplasty and stenting of lower extremity vessels — A balloon or a stent of the required size (according to the intrinsic diameter of the affected vessel) is delivered to the affected area, sequential balloon dilatation with exposure of up to 5 minutes or stenting of the vessel is performed. After completion, control angiography is performed with evaluation of the result. Instruments, introdjuncer are removed. Manual compression haemostasis (up to 20 minutes over the puncture site) followed by aseptic pressure dressing on the puncture site for 12 hours with bed rest.
  Arms: Endovascular treatment

SUMMARY:
Endovascular interventions, such as balloon angioplasty and stenting, are commonly used for PAD due to their proven safety and effectiveness. However, traditional treatments for chronic non-healing wounds are often insufficient. Advances in cell biotechnology, particularly fibroblast therapy, show promise for enhancing wound healing, as fibroblasts play a crucial role in tissue repair and inflammation.

This study aims to develop, assess, and evaluate the safety of a combined treatment approach that incorporates fibroblast therapy with existing methods for managing chronic non-healing wounds in PAD patients.

DETAILED DESCRIPTION:
Chronic obliterative diseases of the lower extremity arteries, or peripheral artery disease (PAD), result from systemic atherosclerosis and affect about 202 million adults globally. This condition, marked by progressive arterial stenosis or occlusion, is associated with significant risk factors such as diabetes, smoking, and hypertension. PAD can lead to symptoms ranging from pain and fatigue to severe complications like non-healing chronic wounds. These wounds impose a substantial economic burden on healthcare systems and significantly impact patients' quality of life.

In some countries, over 2.5 million people suffer from chronic non-healing ulcers, with high rates of recurrence and poor healing outcomes. Managing these wounds is costly, with significant indirect costs due to loss of productivity. Post-amputation survival rates are low, and traditional treatments often fail to fully address the issue.

Endovascular interventions, such as balloon angioplasty and stenting, are preferred for PAD due to their safety and effectiveness. However, current methods for treating chronic non-healing wounds remain insufficient. Recent advancements in cell biotechnology, particularly fibroblast therapy, show promise for improving wound healing. Fibroblasts play a key role in tissue repair and inflammation.

There is a need for more research on the effectiveness of combining fibroblast therapy with existing treatments for chronic non-healing wounds in PAD patients. Addressing this gap could lead to better treatment outcomes and improved quality of life for affected individuals.

The aim of this study is to develop, assess the effectiveness, and evaluate the safety of a combined treatment method for managing chronic non-healing wounds in patients with chronic obliterative disease of the lower extremity arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 75 years inclusive.
2. Patients with a history of confirmed stable intermittent lameness, the symptoms of which have been observed continuously for at least 3 months at the time of randomization.
3. Patients with a diagnosis of PAD (code I 70.2 - I 70.9 according to the International Classification of Diseases, 10th revision [ICD - 10]), confirmed by the results of ultrasound duplex scanning of blood vessels.
4. Patients whose smoking status remained stable for at least 3 months prior to randomization (for smokers).
5. Patients with an ankle - brachial Doppler index value at rest ≤0.9.
6. Patients with a long-term non-healing wound (more than 1 month) and intermittent claudication with a pain-free walking distance of less than 200 meters.
7. Patients who, in the opinion of the investigator, are able to understand and comply with the study requirements.
8. Before starting any examination procedures by the patient or, if applicable, its legal representative, a signed and dated written informed consent form, as well as any necessary processing permissions personal data.

Exclusion Criteria:

1. Acute myocardial infarction (ACS), acute cerebrovascular accident (stroke)
2. Pulmonary embolism (PE)
3. Acute infectious diseases
4. Patients who underwent reconstructive intervention on the arteries of the lower extremities (surgical or intravascular) in the last 3 months before randomization.
5. Patients who underwent major cardiac surgery within 6 months prior to randomization.
6. Patients with congestive heart failure III-IV functional class according to classification of the New York Heart Association.
7. Patients with any other disease that significantly limits physical activity, or any other medical condition that, in the opinion of the investigator, may limit the patient's participation in the study.
8. Patients with mental status disorders
9. Patients with a history of hypersensitivity or allergy to a radiopaque substance, similar drugs or excipients.
10. Patients who are pregnant or breastfeeding, or who plan to become pregnant before participating in this study or during the study, or who intend to become an egg donor within the same period of time.
11. Progression of the underlying and concomitant disease
12. High levels of creatinine and urea in a biochemical blood test (creatinine in women: more than 80.0 µmol / l; men: more than 110.0 µmol / l; ); ( Urea in adults under 60 years of age is more than 8.32 mmol/l, adults over 60 years of age are more than 7.5 mmol/l )
13. Presence of peptic ulcer of the stomach and duodenum (DUD)
14. Patients with total thrombosis of the vessels of the lower extremities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
brachial-shoulder index | 1 day, after 1 month, after 3 month, after 6 month
  The Brachial-Shoulder Index (BSI, ratio) is a diagnostic measure used to assess blood flow and detect potential vascular abnormalities. It is calculated by dividing the systolic blood pressure (mmHg) at the shoulder by the systolic blood pressure (mmHg) at the arm (brachial artery). This index helps evaluate the presence of arterial blockages or compression between the shoulder and the arm, which can indicate peripheral vascular disease or other circulatory issues. A reduced BSI may suggest impaired blood flow (mm/sec) and is useful in diagnosing conditions related to upper limb circulation.

SECONDARY OUTCOMES:
dynamics of wound healing | 1 day, after 1 month, after 3 month, after 6 month
  The dynamics of wound healing refer to the process and progression of tissue repair following an injury. This process involves several key phases:Hemostasis, Inflammation, Proliferation, Maturation. The rate and quality of healing can be influenced by factors such as wound type, underlying health conditions, and treatment methods. Monitoring these dynamics ( in cm^2) helps assess the effectiveness of interventions and guide clinical decisions

OTHER OUTCOMES:
Number of participants | in a month, 3 months, 6 months
  The number of participants in the study will be analyzed.
Analysis of participants' body weight | in a month, 3 months, 6 months
  Participants' body weight will be analyzed
Assessment of the degree of oxygen saturation of the lower extremities | in a month, 3 months, 6 months
  During the study, the oxygen saturation level of the lower extremities will be assessed using a peripheral pulse oximeter. Since ischemia of the extremities affects the oxygen saturation level of the surrounding tissues.
Results of the SF-12 questionnaire | before the tretment, 3 months, 6 months
  Before treatment, then 3 and 6 months after treatment, participants will complete the SF-12 questionnaire, which will take into account the physical condition, mental state and general condition of the participants.
Activity of Daily Living Index - Bartell Index. | before the tretment, 3 months after the treatment, 6 months after the treatment
  The Barthel scale is an ordinal scale used to measure performance in daily living. Each performance element is rated on this scale with a set number of points assigned to each level or ranking. It uses ten variables that describe ADLs and mobility. A higher number is associated with a greater likelihood that you will be able to live at home with a degree of independence after discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Oncology Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No